CLINICAL TRIAL: NCT03295500
Title: On the Cyberknife Dose Fraction of Liver Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: duanxuezhang
Record Dates: First submitted 2017-09-16; First posted 2017-09-28 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: CyberKnife Radiosurgery
Keywords: CyberKnife; hepatocellular; dose fraction; ICG R15

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental Group One: In this group ,the participants receive the dose fraction of 49Gy/7f (BED 83.3Gy) by cyberknife.
  Interventions: Radiation: Dose fraction forms
- Experimental Group Two: In this group ,the participants receive the dose fraction of 54Gy/6f(BED 102.6Gy) by cyberknife.
  Interventions: Radiation: Dose fraction forms
- Control Group: In this group ,the participants receive the dose fraction of 55Gy/5f(115.5Gy) by cyberknife.
  Interventions: Radiation: Dose fraction forms

INTERVENTIONS:
Radiation: Dose fraction forms — The investigators divide the participants randomly into 3 groups by SPSS 19.0.Three groups participants receive the different dose fraction(49Gy/7f,54Gy/6f and 55Gy/5f),which also means different Biologic Equivalent Dose.Through the research,the investigators want to find out the optimum dose fraction method,which makes the treatment safe, effective and personalized.

SUMMARY:
The research aims to the primary hepatic carcinoma patients whose diameter of the single tumor is equal or less than 5cm.By supervising the changes of liver function, Child-Pugh score, ICG-R15 value, secondary reaction, incidence rate of RILD during and after the radiotherapy, meanwhile combining the outcome of the progression of disease and the condition of survival quality, the optimum proposal could be obtained and apply to clinic thus make the treatment safe, effective and personalized.

ELIGIBILITY:
Inclusion Criteria:

* The participants are from 30 to 80 years of age, without gender restriction
* With the hepatopathy background, the diagnosis of primary hepatic carcinoma is confirmed by image examination and laboratory test(the diagnosis criteria is according to the primary hepatic carcinoma rule of diagnosis and treat in 2007)
* The max diameter of single tumor ≤5cm
* Child-Pugh Classification(CPC) A or B
* ECOG score 0 or 1
* Leukocyte is more than 2×109/L and thrombocyte is more than 60×109/L
* Kidney function is normal
* Unsuitable or rejecting other therapies such as resection, liver transplantation etc
* Anticipated lifetime is longer than six months
* The participants who are voluntary comply with the requirements of research
* The participants agree to sign the informed consent.

Exclusion Criteria:

* The metastasis occur outside of liver
* Child-Pugh Classification(CPC)
* The outline of tumor is not confirmed by image examination
* With hepatic or any other abdomen radiotherapy history before
* With severe internal medicine diseases
* Bone marrow haematopoietic function or kidney function is severe failure
* Intractable ascites
* The position of tumor is nearby esophagus, stomach or intestine
* The normal liver volume less than 700 cm3

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to the hepatocellular participants who receive the radiotherapy through different dose fraction by cyberknife.
Sampling Method: Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Local control rate | From date of the participants completing the therapy until the date of first documented progression, assessed up to 36 months.
  Local control illustrates the time from the tumor appearance to progress (the diameter more than or equal to 1.5 times of original) .The ratio of the number of the local control patients to the whole number of patients is local control rate.
Overall survival rate | From date of the participants diagnosed until the date of death from any cause, assessed up to 36 months.
  Overall survival rate means the ratio of the number of patients who are alive to the whole patients after the treatment.

SECONDARY OUTCOMES:
RILD rate | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
  the rate of radiotherapy induced liver disease
Child-Pugh score | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
  By testing the liver function,coagulation function and ascites,we could calculate the Child-Pugh score,which reflect the liver function roundly.
the value of ICG R15 | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
  It means the indocyanine green retention rate at 15 minutes,which reflects the liver reserve.

CONTACTS AND LOCATIONS:
Locations (1):
- CyberKnife, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenmark MH, Cao Y, Wang H, Jackson A, Ben-Josef E, Ten Haken RK, Lawrence TS, Feng M. Estimating functional liver reserve following hepatic irradiation: adaptive normal tissue response models. Radiother Oncol. 2014 Jun;111(3):418-23. doi: 10.1016/j.radonc.2014.04.007. Epub 2014 May 8. PMID 24813090
- [Result] Dewas S, Bibault JE, Mirabel X, Fumagalli I, Kramar A, Jarraya H, Lacornerie T, Dewas-Vautravers C, Lartigau E. Prognostic factors affecting local control of hepatic tumors treated by Stereotactic Body Radiation Therapy. Radiat Oncol. 2012 Oct 10;7:166. doi: 10.1186/1748-717X-7-166. PMID 23050794
- [Result] Goodman BD, Mannina EM, Althouse SK, Maluccio MA, Cardenes HR. Long-term safety and efficacy of stereotactic body radiation therapy for hepatic oligometastases. Pract Radiat Oncol. 2016 Mar-Apr;6(2):86-95. doi: 10.1016/j.prro.2015.10.011. Epub 2015 Oct 23. PMID 26725957
- [Result] Liang P, Huang C, Liang SX, Li YF, Huang SX, Lian ZP, Liu JM, Tang Y, Lu HJ. Effect of CyberKnife stereotactic body radiation therapy for hepatocellular carcinoma on hepatic toxicity. Onco Targets Ther. 2016 Nov 18;9:7169-7175. doi: 10.2147/OTT.S112290. eCollection 2016. PMID 27920555
- [Result] Su TS, Lu HZ, Cheng T, Zhou Y, Huang Y, Gao YC, Tang MY, Jiang HY, Lian ZP, Hou EC, Liang P. Long-term survival analysis in combined transarterial embolization and stereotactic body radiation therapy versus stereotactic body radiation monotherapy for unresectable hepatocellular carcinoma >5 cm. BMC Cancer. 2016 Nov 3;16(1):834. doi: 10.1186/s12885-016-2894-9. PMID 27809890
- [Result] Que J, Kuo HT, Lin LC, Lin KL, Lin CH, Lin YW, Yang CC. Clinical outcomes and prognostic factors of cyberknife stereotactic body radiation therapy for unresectable hepatocellular carcinoma. BMC Cancer. 2016 Jul 12;16:451. doi: 10.1186/s12885-016-2512-x. PMID 27405814
- [Result] Schoenberg M, Khandoga A, Stintzing S, Trumm C, Schiergens TS, Angele M, Op den Winkel M, Werner J, Muacevic A, Rentsch M. CyberKnife Radiosurgery - Value as an Adjunct to Surgical Treatment of HCC? Cureus. 2016 Apr 28;8(4):e591. doi: 10.7759/cureus.591. PMID 27284498
- [Result] Su TS, Liang P, Lu HZ, Liang J, Gao YC, Zhou Y, Huang Y, Tang MY, Liang JN. Stereotactic body radiation therapy for small primary or recurrent hepatocellular carcinoma in 132 Chinese patients. J Surg Oncol. 2016 Feb;113(2):181-7. doi: 10.1002/jso.24128. Epub 2015 Dec 14. PMID 26799260
- [Result] Lo CH, Huang WY, Lin KT, Lin MJ, Lin TP, Jen YM. Repeated stereotactic ablative radiotherapy using CyberKnife for patients with hepatocellular carcinoma. J Gastroenterol Hepatol. 2014 Nov;29(11):1919-25. doi: 10.1111/jgh.12659. PMID 25041220
- [Result] Que JY, Lin LC, Lin KL, Lin CH, Lin YW, Yang CC. The efficacy of stereotactic body radiation therapy on huge hepatocellular carcinoma unsuitable for other local modalities. Radiat Oncol. 2014 May 28;9:120. doi: 10.1186/1748-717X-9-120. PMID 24885086
- [Result] Lo CH, Huang WY, Lee MS, Lin KT, Lin TP, Chang PY, Fan CY, Jen YM. Stereotactic ablative radiotherapy for unresectable hepatocellular carcinoma patients who failed or were unsuitable for transarterial chemoembolization. Eur J Gastroenterol Hepatol. 2014 Mar;26(3):345-52. doi: 10.1097/MEG.0000000000000032. PMID 24384685
- [Result] Bibault JE, Dewas S, Vautravers-Dewas C, Hollebecque A, Jarraya H, Lacornerie T, Lartigau E, Mirabel X. Stereotactic body radiation therapy for hepatocellular carcinoma: prognostic factors of local control, overall survival, and toxicity. PLoS One. 2013 Oct 11;8(10):e77472. doi: 10.1371/journal.pone.0077472. eCollection 2013. PMID 24147002
- [Result] Yoon HI, Koom WS, Lee IJ, Jeong K, Chung Y, Kim JK, Lee KS, Han KH, Seong J. The significance of ICG-R15 in predicting hepatic toxicity in patients receiving radiotherapy for hepatocellular carcinoma. Liver Int. 2012 Aug;32(7):1165-71. doi: 10.1111/j.1478-3231.2012.02784.x. Epub 2012 Mar 21. PMID 22435801
- [Derived] Sun J, Zhang A, Li W, Wang Q, Li D, Zhang D, Duan X. Biologically effective dose (BED) escalation of stereotactic body radiotherapy (SBRT) for hepatocellular carcinoma patients (</=5 cm) with CyberKnife: protocol of study. Radiat Oncol. 2020 Jan 28;15(1):20. doi: 10.1186/s13014-020-1471-1. PMID 31992327